CLINICAL TRIAL: NCT02153580
Title: Phase I Study to Evaluate Cellular Immunotherapy Using Memory-Enriched T Cells Lentivirally Transduced to Express a CD19-Specific, Hinge-Optimized, CD28-Costimulatory Chimeric Receptor and a Truncated EGFR Following Lymphodepleting Chemotherapy in Adult Patients With CD19+ B-Cell Lymphoproliferative Neoplasms
Brief Title: Cellular Immunotherapy Following Chemotherapy in Treating Patients With Recurrent Non-Hodgkin Lymphomas, Chronic Lymphocytic Leukemia, or B-Cell Prolymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13351; NCI-2014-01168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 114025; 122842; 120574; 111658; 13351/117351; 115691; 13351 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Classic Hodgkin Lymphoma; B-Cell Prolymphocytic Leukemia; High Grade B-Cell Lymphoma, Not Otherwise Specified; Post-Transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Hairy Cell Leukemia; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Prolymphocytic, B-Cell; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Hairy Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Cyclophosphamide; Etoposide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (lymphodepletion, cellular immunotherapy) (Experimental): LYMPHODEPLETING REGIMEN: Patients receive a chemotherapy regimen based on disease type and extent of disease comprising of cyclophosphamide, bendamustine hydrochloride, fludarabine phosphate, etoposide.
  CELLULAR IMMUNOTHERAPY: Beginning 3-10 days later after lymphodepletion, patients receive autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes IV over 10-15 minutes on day 0. Patients with relapsed, residual or progressive disease may receive an optional second infusion of autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes >= 28 days post T cell infusion.
  Disease status: Patients with Non-Hodgkin lymphoma (NHL).
  Interventions: Biological: Autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes; Drug: Bendamustine Hydrochloride; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Fludarabine Phosphate
- Group II (lymphodepletion, cellular immunotherapy) (Experimental): LYMPHODEPLETING REGIMEN: Patients receive a chemotherapy regimen based on disease type and extent of disease comprising of cyclophosphamide, bendamustine hydrochloride, fludarabine phosphate, etoposide.
  CELLULAR IMMUNOTHERAPY: Beginning 3-10 days later after lymphodepletion, patients receive autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes IV over 10-15 minutes on day 0. Patients with relapsed, residual or progressive disease may receive an optional second infusion of autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes >= 28 days post T cell infusion.
  Disease status: Patients with Chronic lymphocytic leukemia (CLL) and/or Prolymphocytic Leukemia (PLL).
  Interventions: Biological: Autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes; Drug: Bendamustine Hydrochloride; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: Autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes — Given IV
  Other Names: CD19R(EQ)28zetaEGFRt+ Tn/mem Cells; CD19R(EQ)28zetaEGFRt+ Tn/Tmem
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Belrapzo; Bendamustin Hydrochloride; Bendeka; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586

SUMMARY:
This phase I trial studies the side effects and best dose of cellular immunotherapy following chemotherapy in treating patients with non-Hodgkin lymphomas, chronic lymphocytic leukemia, or B-cell prolymphocytic leukemia that has come back. Placing a modified gene into white blood cells may help the body build an immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of adoptive therapy using ex vivo expanded autologous memory T cells (central memory T cells [Tcm] or naive and memory T-cells [Tn/mem]) that are enriched and genetically modified to express a cluster of differentiation (CD)19-specific, hinged optimized, CD28-costimulatory chimeric antigen receptor (CAR) as well as a truncated human epidermal growth factor receptor (EGFR) (CD19R[EQ]28zeta/truncated EGFR [EGFRt]+ Tcm or CD19R[EQ]28zeta/EGFRt+ Tn/mem) shortly following lymphodepletion for adults with recurrent/progressive/residual CD19 + B-cell lymphoproliferative neoplasms (non-Hodgkin lymphoma [NHL], chronic lymphocytic leukemia [CLL]/prolymphocytic leukemia [PLL]) and who are not eligible for or decline City of Hope (COH) Institutional Review Board (IRB) Protocol Number (No.) 13277.

II. To determine the recommended Phase II dose (RP2D) in the two Tn/mem strata (NHL; CLL/PLL).

SECONDARY OBJECTIVE:

I. To study antitumor activity of CD19R(EQ)CD28zeta/EGFRt+Tcm or CD19R[EQ]28zeta/EGFRt+ Tn/mem (e.g., detection of CAR+ T cells, B cells, and tumor burden).

OUTLINE: This is a dose-escalation study of autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing enriched T cells (T-cell infusion). Participants are assigned to 1 of 2 groups based on disease status.

GROUP I (NON-HODGKIN LYMPHOMA [NHL]):

LYMPHODEPLETING REGIMEN: Patients receive a chemotherapy regimen based on disease type and extent of disease comprising of cyclophosphamide, bendamustine hydrochloride, fludarabine phosphate, etoposide.

CELLULAR IMMUNOTHERAPY: Beginning 3-10 days later after lymphodepletion, patients receive autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes IV over 10-15 minutes on day 0. Patients with relapsed, residual or progressive disease may receive an optional second infusion of autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes >= 28 days post T cell infusion.

GROUP II (CHRONIC LYMPHOCYTIC LEUKEMIA [CLL] AND/OR PROLYMPHOCYTIC LEUKEMIA [PLL]):

LYMPHODEPLETING REGIMEN: Patients receive a chemotherapy regimen based on disease type and extent of disease comprising of cyclophosphamide, bendamustine hydrochloride, fludarabine phosphate, etoposide.

CELLULAR IMMUNOTHERAPY: Beginning 3-10 days later after lymphodepletion, patients receive autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes IV over 10-15 minutes on day 0. Patients with relapsed, residual or progressive disease may receive an optional second infusion of autologous CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes >= 28 days post T cell infusion.

After completion of study treatment, patients are followed up at every 2 days for 14 days, weekly for 1 month, monthly for 1 year, and then yearly for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* SCREENING INCLUSION CRITERIA:
* COH pathology review confirms that research participant's diagnostic material is consistent with recurrent/progressive/residual B cell lymphoproliferative neoplasms as listed below AND the research participant is not eligible for or declines COH IRB Protocol No. 13277; additionally, CD19 positivity must be documented in a pathology report if the research participant previously received CD19-targeted therapy; however, it is not a requirement that the CD19 testing be performed by a COH pathologist

  * Disease stratum 1 (NHL): Unclassifiable high grade lymphoma, mantle cell lymphoma, follicular lymphoma, diffuse large B-cell lymphoma (DLBCL) and all its subtypes, Burkitt lymphoma (BL), marginal zone B-cell lymphoma, hairy cell leukemia, lymphoplasmacytic lymphoma, B cell lymphoma unclassifiable with features intermediate between DLBCL and BL, B cell lymphoma unclassifiable with features intermediate between DLBCL and classical Hodgkin lymphoma, and those research participants who either declined or were not eligible for COH IRB Protocol No. 13277, or who collected autologous T cells for COH IRB Protocol No. 13277 but then became ineligible for autologous hematopoietic stem cell transplant (HSCT) or participants who have relapsed following prior T cell therapy on either COH IRB Protocol No. 09174 or 12224 may be enrolled on this study
  * Disease stratum 2 (CLL/PLL/SLL): chronic lymphocytic leukemia (CLL), and B-cell prolymphocytic leukemia (PLL), and small lymphocytic lymphoma (SLL)
* Karnofsky performance status (KPS) of >= 70%
* Life expectancy >= 16 weeks at time of screening
* The effects of CD19R(EQ)28zeta/EGFRt+ TCM or CD19R(EQ)28zeta/EGFRt+ TN/MEM on the developing fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent

  * Note: For research participants who do not speak English, a short form consent may be used with a COH certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed; however, the research participant is allowed to proceed with lymphodepletion and T cell infusion only after the translated full consent form is signed
* PROTOCOL-SPECIFIC CRITERIA:
* COH pathology review confirms that research participant's diagnostic material is consistent with a lymphoproliferative B-cell neoplasm
* Documentation of recurrence/progression/residual disease following prior therapy
* Negative serum pregnancy test for women of childbearing potential
* A pretreatment creatinine clearance (CrCl) of >= 60 mL/minute (min), calculated by Cockcroft Gault
* Patients must have a serum bilirubin =< 2.0 mg/dl
* Patients must have an alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 times the institutional upper limits of normal
* Ejection fraction measured by echocardiogram or multi gated acquisition scan (MUGA) > 45% (evaluation within 6 weeks of screening does not need to be repeated)
* ELIGIBILITY TO PROCEED WITH PERIPHERAL BLOOD MONONUCLEAR CELL (PBMC) COLLECTION
* Research participant must have appropriate venous access
* Research participant must be at least 2 weeks from having received the last dose of immunosuppressant medications (e.g. calcineurin inhibitors, methotrexate, immunosuppressive antibodies, etc)
* The last dose of prior chemotherapy, immunotherapy or radiation must be at least 2 weeks before the leukapheresis procedure
* The last dose of cytotoxic chemotherapeutic agents that are not considered lymphotoxic must be at least one week before the leukapheresis procedure; oral chemotherapeutic agents, including lenalidomide and ibrutinib, are allowed if at least 3 half-lives have elapsed prior to leukapheresis
* The last dose of lymphotoxic chemotherapeutic agents (e.g. cyclophosphamide, ifosofamide, bendamustine, etc) must be at least 2 weeks before the leukapheresis procedure
* The last dose of investigational agents must be at least 2 weeks before leukapheresis procedure unless no response or disease progression is documented on the experimental therapy and at least 3 half-lives must have elapsed prior to leukapheresis
* Note: exceptions may be made at the discretion of the principal investigator (PI)/study team
* ELIGIBILITY TO UNDERGO LYMPHODEPLETION:
* Research participant has a released cryopreserved T cell product for T cell infusions on approximately day 0
* Research participant must be at least 2 weeks out from having received the last dose of investigational agent
* The last dose of cytotoxic chemotherapeutic agents that are not considered lymphotoxic must be at least one week before lymphodepletion; oral chemotherapeutic agents, including lenalidomide and ibrutinib, are allowed if at least 3 half-lives have elapsed prior to lymphodepletion
* The last dose of lymphotoxic chemotherapeutic agents (e.g. cyclophosphamide, ifosofamide, bendamustine, etc) must be at least 2 weeks before lymphodepletion
* Toxicity related to prior therapy must either have returned to =< grade 3, baseline, or deemed irreversible
* KPS >= 70%
* Participants of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after T cell infusion
* Absolute neutrophil count (ANC) > 0.75
* Platelets > 50 K without growth factor or transfusion support for a week at least
* Not requiring supplemental oxygen or mechanical ventilation, oxygen saturation 90% or higher on room air
* Not requiring pressor support, not having symptomatic cardiac arrhythmias
* Preservation of renal function, serum creatinine did NOT increase by more than 2 fold above the normal range
* Total bilirubin =< 2.0 mg/dL
* Research participant without clinically significant encephalopathy/new focal deficits
* No clinical evidence of uncontrolled active infectious process
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): Research participant has completed prescribed lymphodepletion
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): Not requiring supplemental oxygen or mechanical ventilation, oxygen saturation 90% or higher on room air
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): Not requiring pressor support, not having symptomatic cardiac arrhythmias
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): Preservation of renal function, serum creatinine did NOT increase by more than 2 fold above the normal range
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): Total bilirubin =< 2.0 mg/dL
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): Research participant without clinically significant encephalopathy/new focal deficits
* (ELIGIBILITY CRITERIA AT TIME OF INFUSION OF GENETICALLY MODIFIED AUTOLOGOUS T CELLS): No clinical evidence of uncontrolled active infectious process

Exclusion Criteria:

* SCREENING EXCLUSION CRITERIA:
* Research participants who received memory-enriched CD19R(EQ):CD28:zeta/EGFRt+ on IRB#13277
* Research participants with any uncontrolled illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements
* Research participants with known active hepatitis B or C infection; research participants who are human immunodeficiency virus (HIV) seropositive based on testing performed within 4 weeks of screening; research participants with any signs of symptoms of active infection, positive blood cultures or radiological evidence of infections
* Research participants with presence of other active malignancy; however, research participants with history of prior malignancy treated within 2 years with curative intent and in a complete remission are eligible
* Pregnant and lactating women
* STUDY-SPECIFIC EXCLUSIONS:
* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I study
* Research participants with precursor B-cell acute lymphoblastic leukemia/lymphoma or plasma cell dyscrasias
* Any known contraindications to cyclophosphamide, fludarabine, etoposide, bendamustine, cetuximab or tocilizumab
* Dependence on corticosteroids

  * Steroid dependence can be defined as a medical need to be greater than 5 mg of prednisone (or equivalent doses of other systemic steroids) a day, chronically; higher doses need to be avoided for at least 3 days prior to leukapheresis and, again, for at least 3 days prior to T cell infusion and up to at least 3 months after T cell infusion unless medically indicated to treat a new toxicity
  * Note: topical and inhaled corticosteroids in standard doses and physiologic replacement for subjects with adrenal insufficiency are allowed
* Active autoimmune disease requiring systemic immunosuppressive therapy
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile of T-cell infusion as defined by all toxicities associated with T cells at the probably or definite levels | Up to 15 years
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (v4.0) and modified cytokine release syndrome grading as applicable. Tables will summarize all toxicities and side effects by dose, time post treatment (first 28 days, days 29-60, 61-100, >100 days), organ and severity.
Dose-limiting toxicity rate at the recommended phase II dose assessed using CTCAE v4.0 | Up to 28 days
  Rates and associated 95% Clopper and Pearson binomial confidence limits will be estimated.

SECONDARY OUTCOMES:
Detection of transferred T cells in the circulation for at least 28 days by quantitative-polymerase chain reaction | 28 days
  Rates and associated 95% Clopper and Pearson binomial confidence limits will be estimated.
Disease response by physical exam, lab data, radiographic imaging and, in the case of stratum 2 (chronic lymphocytic leukemia/prolymphocytic leukemia) and leukemic phase non-Hodgkin lymphoma patients by flow cytometry and bone marrow biopsy | Up to 15 years
  Rates and associated 95% Clopper and Pearson binomial confidence limits will be estimated.
CD19 B cell aplasia/immunoglobulin G levels | Up to 15 years
  Normal CD19+ B cell levels and immunoglobulin G levels will be reported over the study period using both descriptive statistics and graphical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Siddiqi, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

REFERENCES:
- [Derived] Siddiqi T, Wang X, Blanchard MS, Wagner JR, Popplewell LL, Budde LE, Stiller TL, Clark MC, Lim L, Vyas V, Brown CE, Forman SJ. CD19-directed CAR T-cell therapy for treatment of primary CNS lymphoma. Blood Adv. 2021 Oct 26;5(20):4059-4063. doi: 10.1182/bloodadvances.2020004106. PMID 34492703